CLINICAL TRIAL: NCT04127409
Title: A Study of the Absorption, Distribution and Cardiovascular Benefits for Humans of Eating Chicken-meat and Eggs Enriched With Omega-3 PUFAs Over a 6-month Period
Brief Title: Impacts of Omega-3-PUFA Enriched Chicken-meat and Eggs in Healthy Humans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alice Stanton (Other)
Collaborators: Devenish Nutrition, Belfast, United Kingdom. (Unknown); Beaumont Hospital (Other); University College Dublin (Other)
Responsible Party: Sponsor-Investigator, Alice Stanton, Professor of Cardiovascular Therapeutics, Royal College of Surgeons, Ireland
Organization: Royal College of Surgeons, Ireland (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: GR15-0981
Record Dates: First submitted 2019-10-06; First posted 2019-10-15 (Actual); Last update posted 2023-11-14 (Actual); Status verified 2023-11

CONDITIONS: Healthy Diet
Keywords: Omega-3 Polyunsaturated Fatty Acids

STUDY DESIGN:
Intervention Model Description: This will be a controlled, double-blind randomized study. Using a 2X2 factorial design, 160 participants will be randomized to eat at least three portions/week of omega-3-PUFA enriched (or control) chicken-meat, and to eat at least three omega-3-PUFA enriched (or control) eggs/week, for 6 months.
  Numbers in each treatment group are indicated below; Control chicken-meat & Control Eggs (n=40) Control chicken-meat & Omega-3 PUFA enriched Eggs (n=40) Omega-3 PUFA enriched chicken-meat & Control Eggs (n=40) Omega-3 PUFA enriched chicken-meat & Omega-3 PUFA enriched Eggs (n=40)
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Randomisation and masking The randomisation schedule was computer generated. Separate sealed opaque envelopes were prepared for male and female participants. All investigators involved in participant recruitment, data collection and entry, sample collection, processing and analysis, will be masked to the randomisation groups until data entry is completed and the database is locked.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control Chicken-meat & Control Eggs (Placebo Comparator): Participants will be provided with control chicken-meat and control eggs, and will be requested to eat at least three portions/week of the control chicken-meat, and to eat at least three control eggs/week, for 6 months.
  Interventions: Other: Control Chicken-meat; Other: Control Eggs
- Control Chicken-meat & Omega-3 Eggs (Experimental): Participants will be provided with control chicken-meat and omega-3-PUFA enriched eggs, and will be requested to eat at least three portions/week of the control chicken-meat, and to eat at least three omega-3-enriched eggs/week, for 6 months.
  Interventions: Other: Control Chicken-meat; Other: Omega-3PUFA Enriched Eggs
- Omega-3 Chicken-meat & Control Eggs (Experimental): Participants will be provided with omega-3-PUFA enriched chicken-meat and control eggs, and will be requested to eat at least three portions/week of the omega-3-PUFA enriched chicken-meat, and to eat at least three control eggs/week, for 6 months.
  Interventions: Other: Control Eggs; Other: Omega-3-PUFA Enriched Chicken-meat
- Omega-3 Chicken-meat & Omega-3 Eggs (Experimental): Participants will be provided with omega-3-PUFA enriched chicken-meat and omega-3-PUFA enriched eggs, and will be requested to eat at least three portions/week of the omega-3-PUFA enriched chicken-meat, and to eat at least three omega-3-PUFA enriched eggs/week, for 6 months.
  Interventions: Other: Omega-3-PUFA Enriched Chicken-meat; Other: Omega-3PUFA Enriched Eggs

INTERVENTIONS:
Other: Control Chicken-meat
  Arms: Control Chicken-meat & Control Eggs; Control Chicken-meat & Omega-3 Eggs
Other: Control Eggs
  Arms: Control Chicken-meat & Control Eggs; Omega-3 Chicken-meat & Control Eggs
Other: Omega-3-PUFA Enriched Chicken-meat
  Arms: Omega-3 Chicken-meat & Control Eggs; Omega-3 Chicken-meat & Omega-3 Eggs
Other: Omega-3PUFA Enriched Eggs
  Arms: Control Chicken-meat & Omega-3 Eggs; Omega-3 Chicken-meat & Omega-3 Eggs

SUMMARY:
Eating oily fish containing long chain seafood-derived omega-3 polyunsaturated fatty acids (PUFAs) protects against heart attacks and strokes. Hence most national and international guidelines now recommend that adults eat at least 2 servings per week of oily fish. However uptake of these recommendations is poor - many people do not eat seafood at all. A number of factors probably contribute to this poor compliance with guidelines; limited availability and costs of oily fish; distaste for oily fish; and concern about toxins in such fish. An Irish company, Devenish Nutrition, offers a possible alternative solution - by feeding omega-3 PUFA-enriched feeds to chicken, Devenish Nutrition have demonstrated that the resultant chicken meat and eggs are enriched in omega-3 PUFAs. A recently completed small study, with 30 participants, showed that 5 weeks of eating omega-3 PUFA enriched chicken resulted in increased blood levels of omega-3 PUFAs. There were also beneficial effects on blood pressure and on platelet stickiness. This study will be larger (including 160 participants) and longer in duration (6 months). It will be a double-blind, controlled, randomized study. This will allow testing whether eating omega-3 PUFA enriched chicken-meat regularly over a 6 month period, results in even greater increments in blood levels of omega-3 PUFAs, and in greater beneficial effects on cardiovascular risk factors. Beneficial effects of eating omega-3 PUFA enriched eggs will also be assessed.

DETAILED DESCRIPTION:
BACKGROUND

There are four long chain omega-3 polyunsaturated fatty acids (PUFAs). Alpha-linolenic acid (ALA 18:3n-3) is found in plants. However the remaining three omega-3 PUFAs, which are longer and more unsaturated (Eicosapentaenoic acid, EPA 20:5n-3, Docosapentaenoic acid, DPA 22:5n-3, and Docosahexaenoic acid, DHA 22:6n-3), are in large part found in oily seafood

Consumption of oily fish, and of long chain seafood-derived omega-3 polyunsaturated fatty acids (PUFAs), has been strongly and consistently associated with reduced cardiovascular morbidity and mortality. In a 2011 "State of the Art Paper" Mozaffarian and colleagues concluded that "current data provide strong concordant evidence that long chain (seafood) n-3 PUFA are bioactive compounds that reduce risk of cardiac death".

Seafood derived omega-3 PUFAs influence a myriad of molecular pathways including membrane structure, ion channel properties, genetic regulation, hepatic fatty acid metabolism, eicosanoid and inflammatory mediator synthesis. It appears likely that the beneficial effects of omega-3 PUFAs are mediated through downstream effects on a range of cardiovascular risk factors including blood pressure, heart rhythm, lipid levels, inflammation, and lastly thrombotic tendency through effects on platelet function. The omega-3 fatty acid docosahexaenoic acid (DHA) is proven essential to pre and postnatal brain development while eicosapentaenoic acid (EPA) is more influential on behaviour and mood.

Because of the strong evidence of benefits of seafood derived omega-3 PUFAs, most national and international guidelines now recommend that adults eat at least 2 servings/week of oily fish (>250 mg/day of long-chain omega-3 PUFAs). However uptake of these recommendations is poor - many people do not consume seafood at all, and approximately one-half of U.S adults consume <60 mg/day of EPA+DHA. A number of factors probably contribute to this poor compliance; limited availability and costs of oily fish; distaste for oily fish; and concern about toxins in such fish including methylmercury, polychlorinated biphenyls and dioxins.

An Irish company, Devenish Nutrition, offers a possible alternative solution - by feeding algae derived omega-3 PUFAs enriched feeds to broiler chicken, Devenish Nutrition have demonstrated that the resultant chicken meat is enriched in EPA, DPA and DHA. Furthermore there was no detrimental effect to bird performance or on taste. Omega-3 enriched eggs are currently commercially available (Skea Egg Farms Ltd, Dungannon, Tyrone), and are produced in a similar fashion, through feeding omega-3 PUFAs enriched feeds to hens.

In a just completed pilot study, portions of omega-3 PUFA enriched chicken-meat were eaten, three times weekly for five weeks, by 30 healthy human volunteers. Plasma levels of the 3 seafood derived omega-3 PUFAs increased from 82 ug/g at baseline to 93 ug/g at five weeks (12% increment, p=0.006), and the red cell omega-3 index (sum of EPA and DHA expressed as percentage of total fatty acids in erythrocyte membranes) increased from 4.9% to 5.1% (p = ns). At 5 weeks, two secondary end-points, blood pressure (BP) and platelet reactivity, had declined significantly in the 30 healthy volunteers - clinic systolic BP reduced from 116 to 113 mmHg (p = 0.014), and urinary thromboxane reduced from 1435 to 1024 pg/mg creatinine (p = 0.037).

In this double-blind, controlled, randomized study, the investigators intend to test whether eating of omega-3 PUFA enriched chicken-meat over a 6 month period, results in greater increments in plasma and red cell levels of omega-3 PUFAs, and in greater beneficial effects on cardiovascular risk factors and on cognitive function and mood. In a second limb to this study the investigators will test for additional beneficial effects in humans of consumption of omega-3 PUFA enriched eggs.

The red cell omega-3 index was chosen as the primary outcome for this study, because of its lessor variability over time compared to plasma values, and because of its proven correlation with EPA and DHA levels in human cardiac tissue, and in multiple relevant organs in animal models.

STUDY AIMS AND OBJECTIVES

The two co-primary objectives are to test whether;

* The consumption of 3 servings of omega-3 PUFA-enriched chicken-meat per week, over a 6 month period, results in measurably higher red cell levels of EPA and DHA.
* The consumption of 3 omega-3 enriched eggs per week, over a 6 month period, results in measurably higher red cell levels of EPA and DHA.

Secondary objectives include the evaluation of:

* Whether the consumption of 3 servings of omega-3 PUFA-enriched chicken-meat per week, over a 6 month period, results in measurably higher plasma levels of EPA and DHA.
* Whether the consumption of 3 omega-3 enriched eggs per week, over a 6 month period, results in measurably higher plasma levels of EPA and DHA.
* Whether the consumption of 3 servings of omega-3 PUFA-enriched chicken-meat per week, over a 6 month period, reduces BP, heart rate, lipid levels, inflammation and/or thrombotic tendencies.
* Whether the consumption of 3 omega-3 enriched eggs per week, over a 6 month period, reduces BP, heart rate, lipid levels, inflammation and/or thrombotic tendencies.
* Whether the consumption of 3 servings of omega-3 PUFA-enriched chicken-meat per week, over a 6 month period, results in improved cognitive function and/or mood.
* Whether the consumption of 3 omega-3 enriched eggs per week, over a 6 month period, results in improved cognitive function and/or mood.

STUDY PARTICIPANTS

160 participants will be recruited to the study through hospital out-patient departments, general practices, and by public advertisement by 2 clinical sites in Dublin, Beaumont and Connolly Hospitals, both of whom are part of the RCSI Teaching Hospital Network Academic Health Centre.

STUDY DESIGN

This will be a controlled, double-blind randomised study. Using a 2X2 factorial design, 160 healthy participants will be randomised to eat at least 3 portions/week of omega-3-PUFA enriched (or control) chicken-meat, and to eat at least 3 omega-3-PUFA enriched (or Control) eggs/week, for 6 months

STUDY CONDUCT

Prior to recruitment to the study, potential participants will be given comprehensive information about the study, unlimited time to study this written information, and all questions will be answered by a study investigator. If the potential participant is satisfied with this information, and wishes to participate, written informed consent will be taken.

At the screening visit, a comprehensive lifestyle and medical history will be taken. A food frequency questionnaire will be completed to capture food intake over the previous year. Clinic and ambulatory blood pressure and heart rate will also be measured, as will height, weight, body mass index, and waist circumference. Finally, assessment of cognitive function and mood will be carried out by a battery of tests. A fasting blood sample will be taken to allow measurement of plasma and red cell levels of EPA and DHA, full blood count (platelet count), renal function, liver function, plasma lipid levels, inflammation (high sensitivity C-reactive protein), platelet function (platelet aggregation and serum thromboxane), and DNA extraction. Urine sampling will also occur to allow assessment of platelet turnover (urinary thromboxane/creatinine ratio), and renal function (microalbuminuria).

After all screening assessments have been completed, and if all inclusion and exclusion criteria are satisfied, participants will be randomized to eating omega-3 PUFA enriched chicken-meat or control chicken-meat, and to omega-3 PUFA enriched eggs or control eggs, for the 6 month period. Randomization will be stratified according to gender.

Omega-3 PUFA enriched chicken (whole chickens, breasts, thighs, drums and wings) and eggs, or the appropriate control chicken and control eggs, will be delivered to the homes of study participants at regular intervals (weekly or two-weekly), so that both they, and up to four family members, will be able to eat at least 3 servings per week of chicken meat, and at least 3 eggs weekly over the 6 month study period. The chicken-meat will be delivered frozen, and the eggs will be delivered refrigerated.

Participants will be asked to avoid the taking of omega-3 PUFA supplements, antihypertensives, lipid lowering therapy, antiplatelet therapy such as aspirin, or any non-steroidal anti-inflammatory drugs (nurofen, indomethacin, diclofenac etc) for the duration of the study. If an analgesic is needed paracetamol may be used.

Participants will be asked to fast, not drink tea or coffee, not smoke and not engage in intense exercise from midnight (minimum 8 hours) prior to the screening (baseline) visit, and prior to the 3 and 6 month visits. Participants may drink water and take essential medications on these mornings. At both the 3 month and the 6 month (final) visit, all baseline assessments will be repeated. At months 1,2,4 and 5 a telephone call will be made to check on participant well-being (absence of adverse events), and on compliance with diet.

STATISTICAL ANALYSIS

Standard summary statistics (mean, standard deviation, median, range, %) will be used to describe baseline characteristics of the participants.

Changes in both the primary and the secondary end-points, at 3 and 6 months from baseline, with consumption of omega-3 enriched chicken-meat and eggs, will be compared to the changes recorded with consumption of control chicken-meat and eggs, using two-way ANOVA.

SAMPLE SIZE CONSIDERATIONS

The primary objective of this study is to test whether the consumption of 3 servings per week of omega-3 PUFA-enriched chicken-meat and/or the consumption of 3 omega-3 PUFA enriched eggs, over a 6 month period results in measurably higher red levels of EPA and DHA (red cell omega-3 index). From the recently completed pilot study, wherein 30 healthy community dwelling subjects ate three servings per week of omega-3-PUFA enriched chicken meat for 5 weeks, the baseline omega-3 index was 4.93% (standard deviation 1.11%). This increased to 5.12% (1.18%) after 5 weeks. The mean difference was 0.19% (0.44%). In order to achieve a power of 95% to detect a difference of 1% in the omega-3 index between those eating control and enriched chicken-meat, and between those eating control and enriched eggs, at a 2-sided-level of 0.05, a sample size of 132 participants is required. To allow for potential losses to follow-up, enrollment of 160 participants is planned.

ELIGIBILITY:
Inclusion Criteria:

* Adults (≥ 18 years)
* Able to give informed consent

Exclusion Criteria:

* Previous diagnosis of significant cardiovascular disease (myocardial infarction, coronary intervention, or stroke).
* Currently prescribed anti-hypertensive, lipid lowering, anti-platelet therapy or non-steroidal anti-inflammatory drugs.
* Discovery of sustained hypertension (Daytime BP average > 140/90), and/or significant dyslipidaemia (Fasting LDL Cholesterol > 4mmol/l or Triglycerides > 4mmol/) at the baseline assessments.
* Currently regularly taking Omega-3 PUFA supplements.
* Any known, unresolved history of drug use or alcohol dependency, lack of ability to comprehend or follow instructions, or unlikely or unable to comply with study follow-up requirements
* Any serious medical condition that may adversely affect the patient's safety, limit the subject's ability to participate in the study, comply with follow-up requirements or impact the scientific integrity of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2015-02-01 (Actual); Primary Completion 2018-08-27 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Red Cell Omega-3 Index | 6 months
  Sum of EPA and DHA expressed as percentage of total fatty acids in erythrocyte membranes

SECONDARY OUTCOMES:
Red Cell Omega-3 Index | 3 months
  Sum of EPA and DHA expressed as percentage of total fatty acids in erythrocyte membranes
Plasma levels of EPA and DHA | 3 and 6 months
  Sum of plasma levels of EPA and DHA (microgram/gram)
Systolic blood pressure | 3 and 6 months
  Mean 24-hour ambulatory systolic blood pressure (mmHg)
Diastolic blood pressure | 3 and 6 months
  Mean 24-hour ambulatory diastolic blood pressure (mmHg)
Heart rate | 3 and 6 months
  Mean 24-hour ambulatory heart rate (beats/minute)
Inflammation | 3 and 6 months
  High-sensitivity C-reactive protein (mg/L)
Thrombotic tendency 1 | 3 and 6 months
  Urinary thromboxane/creatinine ratio (pg/mg creatinine)
Thrombotic tendency 2 | 3 and 6 months
  Platelet count (number/L)
Global cognition | 6 months
  Full-Scale IQ as measured by the WASI II
Executive Function | 6 months
  (Z Verbal Fluency (Letter Fluency) + Z Verbal Fluency (Category Fluency) + Z Verbal Fluency (Switching Fluency) - Z Trail Making Test (Number Letter Switching - [(Number Sequencing + Letter Sequencing)/2]) -Z Colour Word Interference (Inhibition - [(Colour Naming + Word Reading)/2]) - Z Colour Word Interference (Inhibition Switching - [(Colour Naming + Word Reading)/2]))/ 6
Verbal Memory | 6 months
  (Z Word List (Immediate Recall) + Z Word List (Delayed Recall) + Z Word List (Recognition) + Z Logical Memory (Immediate Recall) + Z Logical Memory (Delayed Recall) + Z Logical Memory (Recognition) ) /6
Visual Memory | 6 months
  (Z Complex Figure (Immediate Recall) + Z Complex Figure (Delayed Recall))/2
Information Processing Speed | 6 months
  (Z Trail Making Test (Visual Scanning) + Z Trail Making Test (Number Sequencing) + Z Trail Making Test (Letter Sequencing) + Z Colour Word Interference (Colour naming) + Z Colour Word Interference (Word Reading)) /5) * - 1
Psychomotor Speed | 6 months
  (Z Finger Tapping (Dominant Hand) + Z Finger Tapping (Non-Dominant Hand)) /2
Mood | 6 months
  Hospital Anxiety and Depression Scale

CONTACTS AND LOCATIONS:
Overall Officials: Alice V Stanton, MB PhD, Principal Investigator — Royal College of Surgeons in Ireland
Locations (1):
- Royal College of Surgeons at Beaumont Hospital, Dublin, Ireland

IPD SHARING:
Plan to Share IPD: Yes
All de-identified individual participant data that underlie the results in a publication, and applicable supporting clinical trial documents, may be available upon request.
Supporting Information: Study Protocol, ICF, CSR
Time Frame: 6 months after the primary results have been published
Access Criteria: Formal request from qualified scientific and medical researchers will be considered. Access must be consistent with the principle of safeguarding study participants' privacy and consistent with provision of informed consent